CLINICAL TRIAL: NCT02696174
Title: Effectiveness of A Health Microinsurance Scheme in Improving Health Equity and Clinical Outcomes for Private Primary Care in Kuala Lumpur, Malaysia
Brief Title: Effectiveness of A Health Microinsurance Scheme for Private Primary Care in Malaysia
Acronym: HMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Muralllitharan Munisamy, PhD Research Fellow, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRR 29311
Record Dates: First submitted 2016-02-22; First posted 2016-03-02 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Health Care Quality, Access, and Evaluation; Insurance, Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health Microinsurance Scheme (Experimental): Households owning the HMI package, entitling them to visit and receive treatment from the selected primary care clinic
  Interventions: Other: HMI
- Out-Of-Pocket (No Intervention): Households who visit the selected primary care clinic, but pay by Out-Of-Pocket

INTERVENTIONS:
Other: HMI — A defined priced package of primary care services, including investigation and treatment such as procedures and medication, available at a selected clinic for 6 months
  Other Names: Health Microinsurance Scheme
  Arms: Health Microinsurance Scheme

SUMMARY:
This is the Phase 3 of a 3 phase study to determine the feasibility, acceptability and effectiveness of a health microinsurance scheme in improving health equity and clinical outcomes for private primary care (PPC) in Kuala Lumpur, Malaysia. This two-arm, pre-post, quasi-experimental trial consisted of utilizing a HMI scheme (experimental clinic) and normal OOP payments (control clinic) for 6 months. The HMI scheme enabled subscribed households to access a defined benefit package at a selected PPC for treatment and follow-up.

DETAILED DESCRIPTION:
This will be a quasi-experimental study designed to determine the effectiveness of a community health microinsurance scheme (HMI) in private primary care clinics in Malaysia via a pre-post study of an experimental and control clinic. A proposed HMI scheme, whose price and benefit package have been defined through the earlier Phases 1 and 2, will be accessible to subscribed households at the experimental clinic, while the control clinic has subscribed patients paying as per normal practise, which is by Out-Of-Pocket payment. The HMI scheme enabled subscribers to visit the selected clinic chosen for any form of primary care diagnosis, treatment and follow-up. Both the clinics are located in the Jalan Ipoh area, a suburb of Kuala Lumpur, and have common sociodemographic characteristics. A pre-intervention questionnaire will aim to capture health seeking behaviour, delay in seeking medical care, monthly health expenditure and improvements in clinical outcome (assessed by clinical test results). After six months, a post-intervention questionnaire is administered again to the respondents which then allows assessment of the outcome variables.

ELIGIBILITY:
Inclusion Criteria:

1. Households were located in the study area
2. Method of payment to clinic is by out-of-pocket
3. This is household's regular choice of primary care provider.
4. Patient has been seen in the clinic since at least the past two years i.e from before Jan 1, 2014

Exclusion Criteria:

1. Households had members who died in the year 2014.
2. Households had members who were away from this place of residence for work/transferred for more than 1 month in 2014.
3. Households had members who had regular follow-up in public facilities for chronic disease.
4. Households with members who have switched methods of payment in the last year- (e.g newly bought insurance or retired and lost health benefits so paying OOP)
5. Patients who refuse consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Health-seeking behavior | Change from Baseline health seeking behavior at 6 months
  Delays in seeking healthcare (days)
Monthly health expenditure | Change from Baseline Monthly Health Expenditure at 6 months
  How much has been spent for monthly health expenses (in Ringgit Malaysia)

SECONDARY OUTCOMES:
Clinical Outcome of Diabetes Mellitus | Change from Baseline HbA1c at 6 months
  Measurement of HbA1c
Clinical Outcome of Hypertension | Change from Baseline Resting Mean Blood Pressure at 6 months
  Resting mean blood pressure
Clinical outcome of dyslipidemia | Change from Baseline serum cholesterol and LDL at 6 months
  Total serum cholesterol and LDL
Clinical outcome of bronchial Asthma | Change from Baseline spirometry levels at 6 months
  Spirometry levels

CONTACTS AND LOCATIONS:
Overall Officials: Dr Murallitharan Munisamy, Principal Investigator — College of Public Health Sciences Chulalongkorn University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- Available data/document: Study Protocol — https://www.flipdrive.com/site/login — Username: HMI Password: insurance Total protocol FILE named protocol.pdf
- Available data/document: Informed Consent Form — https://www.flipdrive.com/site/login — Username: HMI Password: insurance Patient Information Sheet and Consent forms in English and Bahasa Malaysia
- Available data/document: Questionnaires — https://www.flipdrive.com/site/login — Username: HMI Password: insurance All questionnaires (English) uploaded